CLINICAL TRIAL: NCT01417962
Title: Post Mortem Magnetic Resonance Imaging in the Fetus, Infant and Child: A Comparative Study With Conventional Autopsy
Brief Title: Magnetic Resonance Imaging Autopsy Study
Acronym: MARIAS
Status: Completed | Type: Observational
Sponsor: Thayyil, Sudhin (Individual)
Collaborators: Great Ormond Street Hospital for Children NHS Foundation Trust (Other); University College London Hospitals (Other)
Responsible Party: Principal Investigator, Sudhin Thayyil, Consultant Neonatologist, Thayyil, Sudhin
Other Study IDs: MR07
Record Dates: First submitted 2011-08-13; First posted 2011-08-16 (Estimated); Last update posted 2013-04-22 (Estimated); Status verified 2013-04

CONDITIONS: Stillbirths; Sudden Infant Death
Keywords: Autopsy; MRI; Stillbirths; Neonatal death; Sudden Infant death
MeSH Terms: conditions — Stillbirth; Sudden Infant Death; Perinatal Death

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Fetuses: Still birth and Termination of pregnancies
- Children: Includes Newborns, Infants and Children

SUMMARY:
The aim of this project is to establish whether magnetic resonance (MR) imaging can provide a minimally invasive approach for post-mortem assessment of the fetus, infant and child, with similar detection rates for anomalies and determination of the cause of death.

This will be achieved by acquiring a database of whole-body, post-mortem MR images in approximately 400 fetuses, infants and children, over a 3 years period. Images will be acquired on a dedicated 1.5T research MR scanner. MR images will be reported by an expert group of paediatric radiologists, and compared, in a blinded fashion, with reports from conventional autopsy performed by expert perinatal and paediatric pathologists. Importantly, the post-mortem information will be assessed with reference to the needs of the parents, referring clinicians and HM Coroners. The detection of central nervous system abnormalities will be assessed separately.

The study will be performed across two sites: A dedicated children's hospital (Great Ormond Street Hospital) and a teaching hospital, with large obstetric, fetal and neonatal departments (University College London Hospital), which are linked academically by University College London.

Co-ordination of the project will be managed by a steering committee, which will ensure accurate collation and comparison of the data.

ELIGIBILITY:
Inclusion Criteria:

* Fetuses, newborns and Infants undergoing conventional autopsy

Exclusion Criteria:

* Lack of parental consent

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This study will be performed across two hospital sites: Great Ormond Street Hospital for Children (GOSH) and University College London Hospitals (UCLH). Both of these hospitals are associated with a single academic institution - University College London (UCL). Consecutive fetuses, newborns and children referred for autopsy at these two hospitals will be eligible for recruitment. All recruited cases will have conventional post-mortem MR imaging at 1.5 Tesla and conventional autopsy. CT imaging will be performed in suspected traumatic injuries and skeletal dysplasias.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2007-03; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Number of cases where the cause of death and/or major pathological lesions are detected | 6 weeks
  Conventional autopsy will be considered as the gold standard. The number (%) of cases where post-mortem MR imaging identifies the cause of death and/or major pathological lesions when compared with conventional autopsy will be reported

SECONDARY OUTCOMES:
MR appearance of death-induced artefacts. | 6 weeks
  The common artefacts seen on post-mortem MR imaging will be described
Number of cases where there is a change in ante-mortem diagnosis | 6 weeks
  Number of cases where there is a change in ante-mortem diagnosis following post-mortem MR imaging will be reported

CONTACTS AND LOCATIONS:
Overall Officials: Andrew M Taylor, MD, Principal Investigator — Great Ormond Street Hospital NHS Trust
Locations (2):
- United Kingdom (2):
  - Great Ormond Street Hospital, London
  - University College Hospital, London

REFERENCES:
- [Result] Sebire NJ, Weber MA, Thayyil S, Mushtaq I, Taylor A, Chitty LS. Minimally invasive perinatal autopsies using magnetic resonance imaging and endoscopic postmortem examination ("keyhole autopsy"): feasibility and initial experience. J Matern Fetal Neonatal Med. 2012 May;25(5):513-8. doi: 10.3109/14767058.2011.601368. Epub 2011 Aug 10. PMID 21740313
- [Result] Thayyil S, De Vita E, Sebire NJ, Bainbridge A, Thomas D, Gunny R, Chong K, Lythgoe MF, Golay X, Robertson NJ, Cady EB, Taylor AM. Post-mortem cerebral magnetic resonance imaging T1 and T2 in fetuses, newborns and infants. Eur J Radiol. 2012 Mar;81(3):e232-8. doi: 10.1016/j.ejrad.2011.01.105. Epub 2011 Feb 23. PMID 21349673
- [Result] Thayyil S, Chitty LS, Robertson NJ, Taylor AM, Sebire NJ. Minimally invasive fetal postmortem examination using magnetic resonance imaging and computerised tomography: current evidence and practical issues. Prenat Diagn. 2010 Aug;30(8):713-8. doi: 10.1002/pd.2534. PMID 20661883
- [Result] Thayyil S. Less invasive autopsy: an evidenced based approach. Arch Dis Child. 2011 Jul;96(7):681-7. doi: 10.1136/adc.2009.165704. Epub 2010 Jun 1. PMID 20515965
- [Result] Thayyil S, Chandrasekaran M, Chitty LS, Wade A, Skordis-Worrall J, Bennett-Britton I, Cohen M, Withby E, Sebire NJ, Robertson NJ, Taylor AM. Diagnostic accuracy of post-mortem magnetic resonance imaging in fetuses, children and adults: a systematic review. Eur J Radiol. 2010 Jul;75(1):e142-8. doi: 10.1016/j.ejrad.2009.10.007. Epub 2009 Nov 11. PMID 19910149
- [Result] Thayyil S, Cleary JO, Sebire NJ, Scott RJ, Chong K, Gunny R, Owens CM, Olsen OE, Offiah AC, Parks HG, Chitty LS, Price AN, Yousry TA, Robertson NJ, Lythgoe MF, Taylor AM. Post-mortem examination of human fetuses: a comparison of whole-body high-field MRI at 9.4 T with conventional MRI and invasive autopsy. Lancet. 2009 Aug 8;374(9688):467-75. doi: 10.1016/S0140-6736(09)60913-2. PMID 19665645
- [Result] Thayyil S, Robertson NJ, Scales A, Weber MA, Jacques TS, Sebire NJ, Taylor AM; MaRIAS (Magnetic Resonance Imaging Autopsy Study) Collaborative Group. Prospective parental consent for autopsy research following sudden unexpected childhood deaths: a successful model. Arch Dis Child. 2009 May;94(5):354-8. doi: 10.1136/adc.2008.150904. Epub 2009 Mar 12. PMID 19282335
- [Result] Thayyil S, Schievano S, Robertson NJ, Jones R, Chitty LS, Sebire NJ, Taylor AM; MaRIAS (Magnetic Resonance Imaging Autopsy Study) Collaborative group. A semi-automated method for non-invasive internal organ weight estimation by post-mortem magnetic resonance imaging in fetuses, newborns and children. Eur J Radiol. 2009 Nov;72(2):321-6. doi: 10.1016/j.ejrad.2008.07.013. Epub 2008 Sep 2. PMID 18768277
- [Result] Thayyil S, Robertson NJ, Scales A, Sebire NJ, Taylor AM. Parental consent for research and sudden infant death. Lancet. 2008 Aug 30;372(9640):715. doi: 10.1016/S0140-6736(08)61298-2. No abstract available. PMID 18761215
- [Result] Schievano S, Sebire NJ, Robertson NJ, Taylor AM, Thayyil S. Reconstruction of fetal and infant anatomy using rapid prototyping of post-mortem MR images. Insights Imaging. 2010 Sep;1(4):281-286. doi: 10.1007/s13244-010-0028-5. Epub 2010 Jun 19. PMID 22347922
- [Derived] Arthurs OJ, Thayyil S, Pauliah SS, Jacques TS, Chong WK, Gunny R, Saunders D, Addison S, Lally P, Cady E, Jones R, Norman W, Scott R, Robertson NJ, Wade A, Chitty L, Taylor AM, Sebire NJ; Magnetic Resonance Imaging Autopsy Study (MaRIAS) Collaborative Group. Diagnostic accuracy and limitations of post-mortem MRI for neurological abnormalities in fetuses and children. Clin Radiol. 2015 Aug;70(8):872-80. doi: 10.1016/j.crad.2015.04.008. Epub 2015 Jun 6. PMID 26050535
- [Derived] Arthurs OJ, Thayyil S, Addison S, Wade A, Jones R, Norman W, Scott R, Robertson NJ, Chitty LS, Taylor AM, Sebire NJ, Offiah AC; Magnetic Resonance Imaging Autopsy Study (MaRIAS) Collaborative Group. Diagnostic accuracy of postmortem MRI for musculoskeletal abnormalities in fetuses and children. Prenat Diagn. 2014 Dec;34(13):1254-61. doi: 10.1002/pd.4460. Epub 2014 Aug 6. PMID 25043483
- [Derived] Taylor AM, Sebire NJ, Ashworth MT, Schievano S, Scott RJ, Wade A, Chitty LS, Robertson N, Thayyil S; Magnetic Resonance Imaging Autopsy Study Collaborative Group. Postmortem cardiovascular magnetic resonance imaging in fetuses and children: a masked comparison study with conventional autopsy. Circulation. 2014 May 13;129(19):1937-44. doi: 10.1161/CIRCULATIONAHA.113.005641. Epub 2014 Mar 19. PMID 24647275
- [Derived] Thayyil S, Sebire NJ, Chitty LS, Wade A, Olsen O, Gunny RS, Offiah A, Saunders DE, Owens CM, Chong WK, Robertson NJ, Taylor AM. Post mortem magnetic resonance imaging in the fetus, infant and child: a comparative study with conventional autopsy (MaRIAS Protocol). BMC Pediatr. 2011 Dec 22;11:120. doi: 10.1186/1471-2431-11-120. PMID 22192497